CLINICAL TRIAL: NCT04058769
Title: Software Development for Anesthesiology Guideline Implementation in the Perioperative Course
Brief Title: Software-guided Guideline Implementation in Premedication
Acronym: SGGIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Health Information Management, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 38/19 S-SR
Record Dates: First submitted 2019-08-08; First posted 2019-08-16 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-03

CONDITIONS: Pre-operative Assessment; Adults; Non-cardiac Surgery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Software first (Other): Patients that are pre-operatively assessed first software-guided and then traditional
  Interventions: Device: Premedication Guide
- Traditional (Other): Patients that are first pre-operatively assessed in the traditional way and then with aid of the software
  Interventions: Device: Premedication Guide

INTERVENTIONS:
Device: Premedication Guide — Software with guidelines recommendations for preoperative assessment

SUMMARY:
Aim of the project is the development of a software for implementation of anesthesiology guidelines in the preoperative evaluation. The software bases on the 2014 and 2018 guidelines of the European Society of Anesthesiology (ESA) for the pre-operative evaluation of adults undergoing non-cardiac surgery.

Traditional premedication is compared with the new software-guided premedication by using a cross-over design. 200 patients are included in the study, 100 of which are first evaluated the traditional way and then with the software, 100 patients are treated the other way round. Results of the two premedication methods are compared according to the primary endpoint "correct approval for OP" and the secondary endpoints number of missed apparative examinations, number of unnecessary apparative examinations, time required for premedication, length of hospital stay, mortality and postoperative complications.

DETAILED DESCRIPTION:
Type of study:

Monocentric, prospective cohort study

Procedure for informing and obtaining consent:

Patients who are prepared for surgery in the anesthetic outpatient department or enrolled in the pre-medication list and who meet all inclusion criteria and no exclusion criteria will be identified before the anesthesia consultation. The patients will be informed about the purpose and the course of the study in oral and written form, after which the written consent of the patient will be given before the study-relevant data and examinations are carried out.

Description of the data sources (medical records, questionnaires, etc.):

Data Sources: Patient's medical history, patient history and physical examination, data on standardized Thieme Compliance anesthesia sheets, and existing findings, either external, patient-brought or in-house findings from the SAP. These data are entered into the PDMS. The name of the premedic anesthetist is not relevant for the evaluation and will not be deposited.

Listing / description of the data to be collected:

With the PDMS, all anesthesia-relevant data is collected. These include the history of the patient, current complaints, medication history, physical examination and findings from supplementary equipment examinations. The data of the anonymized control group are extracted exclusively from the PDMS.

Timing (appointments) for the individual study participant:

After the patient has been informed and has consented, after randomization either the premedication as usual with the "old PDMS module" is performed and then a second time with the new software module by another doctor or vice versa, first with the new software and then in the traditional way. This type of cross-over design is done to avoid carry-over effects. The conventional premedicating physician does not know about the patient's participation in the study and makes the decision about the OP release as well as any necessary additional examinations in the usual way and dismisses the patient with the usual pre-hospitalization standard.

The premedication with the new software module is carried out by a doctor who has been trained in it and does not know the result of the first premedication interview. With the help of the new software, the decision on release and possible additional examinations is also made here. The data from the two premedication interviews are stored in xml format in the MRI Data Room and entered in a pseudonymized form in a database. This is done promptly on the day of premedication. A specialist trained in the guidelines, who is blinded to the premedication procedure, compares the results of both premedications. He decides whether the release was correct in both of the above cases or not. If it turns out that the results of both premedications differ and possibly a revision of the premedication document is necessary, unblinding and, if necessary, correction of the premedication document takes place.

Furthermore, the time required for the premedication interview is analyzed as well as the correct arrangement of additional examinations. The secondary outcome parameters are collected using the KIS (clinic information system) and PDMS.

As a comparison population with respect to the secondary endpoints, a conventionally premedicated patient collective, whose anonymized data is extracted from the existing PDMS database, is used in the same period. The endpoint of the comparison is the occurrence of postoperative complications corresponding to a clavia-dindo score of ≥ 3. This corresponds to the events of re-intervention, admission to intensive care unit or death.

Expected end of data collection With hospital discharge, the data collection for the individual patient is completed.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* ASA 3 or 4
* elective surgery
* written informed consent

Exclusion Criteria:

* emergency surgery
* patient not being able to give informed consent
* non-german-speaking patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
correct approval for operation | 1 day
  number of patients that were approved correctly for surgery

SECONDARY OUTCOMES:
missing examinations | 1 day
  number of examinations that were recommended by the guidelines but not applied to the patient
unnecessary examinations | 1 day
  number of examinations that were not recommended by the guidelines but nevertheless applied
mortality | 30 days
  in-hospital mortality
length of hospital stay | 30 days
  length of hospital stay
postoperative complications | 30 days
  postoperative complications assessed by the Clavien-Dindo-Classification (I: no intervention, II: pharmacologic intervention, IIIa:intervention without general anesthesia, IIb: intervention requiring general anesthesia, IV:life-threatening intervention with dysfunction of one organ, IVb: life-threatening intervention with multi-organ dysfunction, V:death

CONTACTS AND LOCATIONS:
Locations (1):
- TU Muenchen, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kagerbauer SM, Wissler J, Andonov DI, Ulm B, Schneider G, Podtschaske AH, Blobner M, Jungwirth B. Implementation of a software-based decision support tool for guideline-appropriate preoperative evaluation: a prospective agreement study. Br J Anaesth. 2024 Sep;133(3):519-529. doi: 10.1016/j.bja.2024.06.001. Epub 2024 Jul 5. PMID 38971713